CLINICAL TRIAL: NCT04583540
Title: Health Status and Quality of Life in Postpartum Women With Placenta Accrete Spectrum.
Brief Title: Quality of Life in Postpartum Women With Placenta Accrete Spectrum.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Beshoy Atef Mounir Rizk, Resident doctor, Assiut University
Other Study IDs: QOL placenta accrete
Record Dates: First submitted 2020-09-23; First posted 2020-10-12 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2020-10

CONDITIONS: Placenta Accrete Spectrum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. The objective of this study is to provide an overview of the core domains (physical,psychological,social) of quality of life and health state in postpartum women after the placenta accrete spectrum.
2. to assess which factors are associated with quality of life and health state domains postpartum.

DETAILED DESCRIPTION:
The morbidly adherent placenta is abnormally adherent placenta to myometrium due to the absence of decidua basalis partially or totally in a way that prevents normal placental separation after delivery.

MAP includes a spectrum classified according to the extend of trophoblastic invasion to myometrium into (accrete, increta, percreta).

The greatest risk factor is previous uterine surgery mostly previous caesarian sections.

In the last decade incidence of placenta accrete spectrum has increased in direct proportion with increased rates of cesarean sections up to 1 per 500 pregnancies.

This rising incidence makes placenta accrete spectrum (PAS)one of the most serious problems in obstetrics with a high rate of complications peripartum and postpartum as well like (peripartum hysterectomy - intestinal injure- bladder injure - ureteral injure - ICU admission- massive blood transfusion) that may affect patients health outcome and their quality of life.

Diagnosis of PAS depends mainly on the history of antepartum hemorrhage and confirmed by the grayscale US with high sensitivity and specificity reaching up to 90%.

Medical service is no longer one-sided evaluated. Patient-centered care is a core in medical service.

Quality of life (QOL) and health status (HS) are important categories of patient-reported outcomes (PROs), in which the patient's perspective is key, and that can be used to assess the impact of current HS and to assess the efficiency of interventions. The difference between these PROs is that where HS refers to self-perceived physical, psychological, and social functioning, QOL also incorporates patients' evaluation of functioning, i.e. (dis)satisfaction with the aspects of life. Since health care is becoming more and more patient-centered, the assessment of the patient's subjective experience is considered to be essential for informed clinical decision-making and health policy. Therefore, research on QOL and HS in postpartum women is increasing, in which multiple contributing factors and interventions are examined.

The WHOQOL is a quality of life assessment developed by the WHOQOL Group with fifteen international field centers, simultaneously, in an attempt to develop a quality of life assessment that would be applicable cross-culturally.

The WHOQOL-Bref scoring assesses four domains of quality of life with 26 items 1_physical health, 2-psychological health, 3- social relationships, 4- environment.

The short form 36 ( SF-36) score is validated quality of life survey with 36 items to assess health outcome and quality of life through eight domains 1- physical functioning (PF), 2-role limitation due to the physical problem ( RP), 3-bodily pain (BP), 4- general health (GH), 5- vitality (VT), 6- social functioning (SF), 7- role limitation due to emotional problem (RE), 8- mental health (MH).

The objective of this research is to assess the quality of life in patients who had placenta accreta spectrum using WHOQOL-BREF scoring and SF-36 quality of life survey

ELIGIBILITY:
Inclusion Criteria:

* 1-Confirmed diagnosis of MAP. 2-Termination of pregnancy after 36 weeks gestation 3-Peripartum hysterectomy for MAP. 4- Complicated CS without hysterectomy 5-Maternal age between 18 and 45 yrs 6-No other medical diseases

Exclusion Criteria:

1. Emergency CS before confirming MAP diagnosis.
2. Preterm delivery (before 36 weeks in case of MAP)
3. .peripartum hysterectomy for any cause other than MAP
4. Other medical diseases that affect the quality of life
5. Postpartum depression.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: All women have confirmed diagnosis of placenta accrete spectrum by Doppler abdominal ultrasound termination of pregnancy by elective cs after fullterm.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess quality of life in patients had placenta accrete spectrum 6-8 weeks postpartum | Baseline
  Use of SF-36 survey to assess quality of life in women had placenta accrete spectrum 6-8 weeks postpartum
patients had placenta accrete spectrum 6-8 weeks postpartum | Baseline
  Use of WHOQOL-bref scoring to assess quality of life in women had placenta accrete spectrum 6-8 weeks postpartum

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Assiut university, Asyut, Egypt